CLINICAL TRIAL: NCT00051636
Title: Randomized, Double-blind, Safety and Efficacy Trial With Intravenous Zoledronic Acid for the Treatment of Paget's Disease of Bone Using Risedronate as a Comparator, Including an Extended Observational Period
Brief Title: Safety and Efficacy Trial With Zoledronic Acid for the Treatment of Paget's Disease of Bone, Including an Extended Observation Period
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CZOL446H2304; ZOL446K2304 (Other: Novartis Pharmaceuticals); NCT00050258 (obsolete NCT alias)
Record Dates: First submitted 2003-01-14; First posted 2003-01-15 (Estimated); Results first posted 2012-05-07 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Paget's Disease of Bone
Keywords: Bisphosphonate; SAP; SAP excess; non-inferiority; therapeutic response; extended observation period
MeSH Terms: conditions — Osteitis Deformans | interventions — Zoledronic Acid; Risedronic Acid; Calcium; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Zoledronic Acid and Placebo to Risedronate (Experimental): Participants received zoledronic acid 5 mg intravenous infusion one dose, 60 days of oral placebo to risedronate, calcium 500 mg twice a day and vitamin D 400 to 1000 international units daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
  Interventions: Drug: Zoledronic Acid; Drug: Placebo to Risedronate; Dietary Supplement: Calcium and Vitamin D
- Risedronate and Placebo to Zoledronic Acid (Active Comparator): Participants received 60 days of oral risedronate 30 mg, one intravenous infusion of placebo to zoledronic acid, calcium 500 mg twice a day and vitamin D 400 to 1000 international units daily during the core period, and received only calcium and vitamin D supplements during the extended observation period.
  Interventions: Drug: Risedronate; Drug: Placebo to Zoledronic Acid; Dietary Supplement: Calcium and Vitamin D

INTERVENTIONS:
Drug: Zoledronic Acid — Zoledronic acid 5 mg in 5 mL of sterile water intravenous infusion.
  Other Names: Reclast, Aclasta
  Arms: Zoledronic Acid and Placebo to Risedronate
Drug: Risedronate — Oral risedronate 30 mg capsules.
  Other Names: Actonel
  Arms: Risedronate and Placebo to Zoledronic Acid
Drug: Placebo to Risedronate — Oral placebo of risedronate capsules.
  Arms: Zoledronic Acid and Placebo to Risedronate
Drug: Placebo to Zoledronic Acid — 5 mL of sterile water one dose intravenous infusion.
  Arms: Risedronate and Placebo to Zoledronic Acid
Dietary Supplement: Calcium and Vitamin D — Calcium and vitamin D supplements were supplied.

SUMMARY:
The core study looked at the effect of Zoledronic Acid given once as an intravenous (i.v.) infusion compared to 60 days of oral Risedronate in patients with Paget's disease of bone. The effect was demonstrated in the reduction of serum alkaline phosphatase (SAP). The extended observation period included participants of the core study who responded to treatment.

ELIGIBILITY:
Inclusion Criteria:

* 30 years or older
* Serum alkaline phosphatase (SAP) 2 times upper limit normal (ULN)
* Confirmed diagnosis of Paget's disease of the bone (by x-ray, magnetic resonance imaging, computerized tomography, radioisotope imaging, etc.).
* 90 days washout calcitonin
* 180 day washout bisphosphonate

Exclusion Criteria:

* Allergic reaction to bisphosphonates
* History of upper gastrointestinal disorders
* History of iritis, uveitis
* Calculated creatinine clearance < 30 ml/min at baseline
* Evidence of vitamin D deficiency

Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2001-01; Primary Completion 2004-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (12):
  - Novartis Investigative Site, Santa Monica, California
  - Novartis Investigative Site, Lakewood, Colorado
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative site, Maywood, Illinois
  - Novartis investigative site, Worcester, Massachusetts
  - Novartis investigative site, Detroit, Michigan
  - Novartis Investigative Site, New York, New York
  - Novartis investigative site, Syracuse, New York
  - Novartis investigative site, Durham, North Carolina
  - Novartis investigative site, Medford, Oregon
  - Novartis investigative site, Providence, Rhode Island
- Australia (6):
  - Novartis Investigative Site, Concord
  - Novartis Investigative Site, Fitzroy
  - Novartis Investigative site, Geelong
  - Novartis Investigative Site, Kogarah
  - Novartis Investigative site, Maroochydore
  - Novartis Investigative site, Nedlands
- Canada (5):
  - Novartis Investigative Site, Calgary
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Montreal
  - Novartis Investigative Site, Ste-Foy
  - Novartis Investigative Site, Toronto
- New Zealand (2):
  - Novartis Investigative site, Auckland
  - Novartis Investigative Site, Christchurch
- Novartis Investigative site, Salamanca, Spain
- United Kingdom (8):
  - Novartis Investigative site, Liverpool
  - Novartis Investigative Site, Manchester
  - Novartis Investigative site, Nottingham
  - Novartis Investigative Site, Oxford
  - Novartis Investigative site, Penarth
  - Novartis investigative site, Pernarth
  - Novartis Investigative Site, Stanmore
  - Novartis Investigative Site, Vale of Glamorgan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 172 participants entered period 1; of these, 127 were identified as treatment responders and entered the extended observation period 2. Responders defined as patient who had ≥75% decrease from baseline in serum alkaline phosphatase (SAP) excess (difference between measured level and midpoint of normal range) or SAP within normal range at 6 months.
Period: Period 1 - Core
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Started | 90 | 82
Completed | 86 | 76
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 0 | 2
Period: Period 2- Extended Observation Period
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Started | 75 | 52
Completed | 5 (Includes patients retreated for Paget's disease and patients discontinued when sponsor ended study) | 22 (Includes patients retreated for Paget's disease)
Not Completed | 70 | 30
Not completed — Lost to Follow-up | 5 | 4
Not completed — withdrew for nonclinical reason | 12 | 7
Not completed — Clinical reasons other than Paget's | 9 | 2
Not completed — Death | 4 | 5
Not completed — Amendment 6 Informed Consent Not Signed | 40 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid | Total
Number analyzed (Participants) | 90 | 82 | 172
Age Continuous [Mean (Standard Deviation); unit: years] | 70.4 (10.25) | 72.1 (9.91) | 71.2 (10.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 21 | 49
  Male | 62 | 61 | 123

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieve Therapeutic Response at 6 Months.
Description: Therapeutic response is defined as a reduction of at least 75% from baseline (Visit 1) in total serum alkaline phosphatase excess (difference between measured level and midpoint to the normal range) or normalization of serum alkaline phosphatase at the end of six months.
Time Frame: 6 months
Population: Modified intent to treat population: all randomized patients with both baseline and at least one post-baseline serum alkaline phosphatase measurement. Missing values at 6 months were imputed using the last post-baseline measurement prior to 6 months.
Measure: Number; unit: participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 88 | 82
participants | 85 | 60

2. Secondary Outcome: Relative Change in Serum Alkaline Phosphatase (SAP) in Units Per Liter (U/L) at Day 28
Description: The percent change in serum alkaline phosphatase from baseline to day 28 was measured.
Time Frame: Baseline and day 28
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and 28 days were included in this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 79 | 79
percent change | -48.8 (11.51) | -28.4 (17.72)

3. Secondary Outcome: Relative Change in Serum C-telopeptide (CTx) in ng/mL at Day 10
Description: The percent change in serum C-telopeptide from baseline to day 10 was measured.
Time Frame: Baseline and day 10
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and day 10 were included in this analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 75 | 72
percent change | -85.4 (18.00) | -36.7 (69.58)

4. Secondary Outcome: Relative Change in Urine Alpha C-telopeptide (α-CTx) in ug/mmol at Day 10
Description: The percent change in urine alpha C-telopeptide from baseline to day 10 was measured.
Time Frame: Baseline and day 10
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 77 | 73
Percent change | -90.3 (13.19) | -29.9 (37.52)

5. Secondary Outcome: Time to First Therapeutic Response
Description: A therapeutic response was defined as a reduction of at least 75% from baseline (Visit 1) in serum alkaline phosphatase excess (difference between measured level and midpoint to the normal range) or normalization of serum alkaline phosphatase.
Time Frame: 182 days
Population: Intent-to-treat population: all randomized patients.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 90 | 82
Days | 64 [61 to 65] | 78 [64 to 178]

6. Secondary Outcome: Number of Patients Who Achieved Serum Alkaline Phosphatase Normalization at Day 28 Relative to Baseline
Description: Normalization of serum alkaline phosphatase occurred if the serum alkaline phosphatase measurement fell within the normal range.
Time Frame: Baseline and day 28
Population: Intent-to-treat population: all randomized patients. Participants with observations at day 28 were included in this analysis.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 88 | 82
Participants | 5 | 0

7. Secondary Outcome: Change in Pain Severity Score
Description: Change in pain severity score from Brief Pain Inventory-Short Form (BPI-SF). This scale values are 0 to 10, a lower score means little to no pain while a higher score means greater pain.
Time Frame: Baseline and day 182
Population: Intent-to-treat population: all randomized patients. Participants with observations at baseline and day 182 were included in this analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 51 | 46
Units on a scale | -0.5 (1.77) | -0.7 (2.22)

8. Secondary Outcome: Change in Pain Interference Score
Description: Change in pain interference score from Brief Pain Inventory-Short Form (BPI-SF). This scale values are 0 to 10, a lower score means little to no pain while a higher score means greater pain.
Time Frame: Baseline and day 182
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 51 | 45
Units on a scale | -0.2 (1.97) | 0.1 (1.72)

9. Secondary Outcome: Number of Participants With a Loss of Therapeutic Response During the Extended Observation Period
Description: Extended observation period. A therapeutic response is defined as a reduction of at least 75% from baseline in serum alkaline phosphatase excess or normalization of serum alkaline phosphatase.
Time Frame: 8 years was the maximum
Population: Extended modified Intent-to-treat population: patients who had at least one serum alkaline phosphatase measurement during the extension period.
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 75 | 52
Participants | 8 [NA to NA] | 29 [368 to NA]

10. Secondary Outcome: Number of Participants With a Partial Disease Relapse During the Extended Observation Period
Description: Extended observation period. A partial disease relapse was defined as an increase in serum alkaline phosphatase >= 50% from the serum alkaline phosphatase measurement at month 6 and at least 1.25 times the upper normal limit.
Time Frame: 8 years was the maximum
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 75 | 52
Participants | 6 [NA to NA] | 26 [547 to NA]

11. Secondary Outcome: Number of Participants With a Disease Relapse During the Extended Observation Period
Description: Extended observation period. A disease relapse was defined as the occurrence of a serum alkaline phosphatase level that was >= 80% of baseline serum alkaline phosphatase value.
Time Frame: 8 years was the maximum
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Number analyzed (Participants) | 75 | 52
Participants | 0 [NA to NA] | 7 [1739 to NA]

ADVERSE EVENTS:
Description: The safety population consisted of all randomized patients who were exposed to study drug.
Arm/Group | Zoledronic Acid and Placebo to Risedronate | Risedronate and Placebo to Zoledronic Acid
Serious Adverse Events (participants affected / at risk) | 5/89 | 8/82
Other Adverse Events (participants affected / at risk) | 71/89 | 58/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid and Placebo to Risedronate (N=89) | Risedronate and Placebo to Zoledronic Acid (N=82)
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Difficulty in walking (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Rigors (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 0 | 1
Cellulitis orbital (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Leg amputation (Surgical and medical procedures) | 1 | 0
Sympathectomy (Surgical and medical procedures) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid and Placebo to Risedronate (N=89) | Risedronate and Placebo to Zoledronic Acid (N=82)
Constipation (Gastrointestinal disorders) | 5 | 6
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Dyspepsia (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 10 | 8
Fatigue (General disorders) | 8 | 5
Influenza like illness (General disorders) | 6 | 4
Oedema peripheral (General disorders) | 5 | 1
Pain (General disorders) | 7 | 5
Pyrexia (General disorders) | 11 | 1
Rigors (General disorders) | 13 | 0
Influenza (Infections and infestations) | 8 | 6
Nasopharyngitis (Infections and infestations) | 8 | 10
Fall (Injury, poisoning and procedural complications) | 8 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 9
Dizziness (Nervous system disorders) | 10 | 3
Headache (Nervous system disorders) | 10 | 11
Lethargy (Nervous system disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.